CLINICAL TRIAL: NCT02229461
Title: A Randomized, Open Label, Parallel Group Study to Investigate the Effects on Serum Thromboxane by the Addition of Naproxen Sodium to Aspirin Therapy Versus Aspirin Therapy Alone
Brief Title: Naproxen Sodium/ASA Platelet Study
Acronym: Kontakt
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15525
Record Dates: First submitted 2014-07-31; First posted 2014-09-01 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Hematology
MeSH Terms: interventions — Naproxen; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- IR ASA co-administered with naproxen sodium (Experimental): Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg once daily (qd) in parallel with naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- IR ASA 30 min after naproxen sodium (Experimental): Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 30 minutes after naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- IR ASA 8 hours after naproxen sodium (Experimental): Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 8 hours after naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- IR ASA only (Active Comparator): Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd. A 3-day IR ASA 81 mg qd Run-Out period was followed.
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- IR ASA 30 min before naproxen sodium (Experimental): Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 30 minutes before naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- IR ASA 30 min after first dose of naproxen sodium bid (Experimental): Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 30 minutes after first dose of naproxen sodium (Aleve, BAY117031) 220 mg, followed by second dose of naproxen sodium 220 mg 12 hours after first dose, for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)

INTERVENTIONS:
Drug: Naproxen Sodium (Aleve, BAY117031) — Naproxen sodium 220 mg qd or bid
  Arms: IR ASA 30 min after first dose of naproxen sodium bid; IR ASA 30 min after naproxen sodium; IR ASA 30 min before naproxen sodium; IR ASA 8 hours after naproxen sodium; IR ASA co-administered with naproxen sodium
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — ASA 81 mg qd

SUMMARY:
To determine if administration of naproxen sodium 220 mg maintains the platelet inhibitory effect of a low dose Immediate Release Aspirin (IR ASA) regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 18 - 70 years of age with a Body Mass Index (BMI) of approximately 18 to 30 kg/m2, and a total body weight > 50 kg (110 lbs)
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Depo-Provera®, or a double barrier and have a negative pregnancy test at Screening and immediately prior to investigational product administration on Day 1 and Day 6. Female subjects of non-childbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the Principal Investigator and the Sponsor
* Be willing and able to participate in all scheduled visits, treatment plan, laboratory tests and other trial procedures according to the protocol
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* History of hypersensitivity or asthma type symptoms with use of aspirin, naproxen sodium and similar pharmacological agents or components of the products
* Females who are pregnant or lactating
* Any disorder of the Aspirin Triad Syndrome (i.e., asthma, rhinitis or nasal polyps), or have chronic urticaria
* Eighteen to twenty years old with a viral infection, with or without fever within one month prior to start of Run-in Period
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, infectious diseases or malignancies
* Any abnormal laboratory value or physical finding that according to the Investigator that may interfere with the interpretation of the study results or be indicative of an underlying disease state
* Have taken any medications including NSAIDs (except acceptable forms of birth control) within 7 days prior to the start of the Run-in Period or throughout the study, unless in the opinion of the Investigator and the Sponsor, the medication will not interfere with the study procedures, data integrity, data interpretation or compromise the safety of the subject
* Have taken antiplatelet or anticoagulant drugs within 30 days prior to start of the Run-in Period or during their participation in the study
* Have donated blood or blood components within 30 days prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Austin, Texas, United States

REFERENCES:
- [Derived] Gurbel PA, Bliden KP, Zhu J, Troullos E, Centofanti R, Jarvis S, Venkataraman P, Tantry US. Thromboxane inhibition during concurrent therapy with low-dose aspirin and over-the-counter naproxen sodium. J Thromb Thrombolysis. 2018 Jan;45(1):18-26. doi: 10.1007/s11239-017-1593-y. PMID 29198079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single site in United States between 16-Feb-2015 (first patient first visit) and 08-May-2015 (last patient last visit).
Pre-assignment Details: Of 117 screened participants in Run-In period, 15 were not randomized into Treatment Period. 2 participants were not randomized because of non-compliance; 3 because of investigator's decision; the other 10 because of other reasons (e.g arachidonic acid-induced platelet aggregation≥20% or pre-randomization elimination of back-up participants).
Groups:
- Group 1-IR ASA Co-administered With Naproxen Sodium: Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg once daily (qd) in parallel with naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
- Group 2-IR ASA 30 Min After Naproxen Sodium: Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 30 minutes after naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
- Group 3-IR ASA 8 Hours After Naproxen Sodium: Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 8 hours after naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
- Group 4-IR ASA Only: Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd. A 3-day IR ASA 81 mg qd Run-Out period was followed.
- Group 5-IR ASA 30 Min Before Naproxen Sodium: Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 30 minutes before naproxen sodium (Aleve, BAY117031) 220 mg qd for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
- Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid: Confirmed eligible participants were randomized to be administered immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg qd 30 minutes after first dose of naproxen sodium (Aleve, BAY117031) 220 mg, followed by second dose of naproxen sodium 220 mg 12 hours after first dose, for 10 consecutive days. A 3-day IR ASA 81 mg qd Run-Out period was followed.
Period: Overall Study
Arm/Group | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid
Started | 17 (Randomized and received treatment) | 17 (Randomized and received treatment) | 17 (Randomized and received treatment) | 17 (Randomized and received treatment) | 17 (Randomized and received treatment) | 17 (Randomized and received treatment)
Completed | 17 | 17 | 17 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Randomized: Fifteen participants were not randomized into Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid | Non-Randomized | Total
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17 | 15 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (8.46) | 31.2 (7.19) | 37.5 (13.41) | 34.2 (8.76) | 38.8 (12.09) | 38.9 (10.62) | 38.2 (13.74) | 37.1 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 6 | 4 | 4 | 7 | 4 | 36
  Male | 10 | 13 | 11 | 13 | 13 | 10 | 11 | 81

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Serum Thromboxane B2 (TXB2) on Day 16 at 24 Hour Post IR ASA 81 mg Administration
Description: Inhibition of serum TXB2 at specified time point was calculated using the percentage of reduction from baseline as follows: Inhibition (%) = 100 × (Baseline Value - Post-baseline Value) / Baseline Value. For primary analysis, the mean and the lower bound of the corresponding one-sided 95% Confidence Interval (CI) were calculated.
Time Frame: At hour 24 on Day 16 post treatment
Population: Percentages are based on the number of participants in the Evaluable Population in each treatment group.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 10 | 15
percentage | 93.09 [91.50 to NA] — One-sided 95% CI | 87.71 [85.51 to NA] — One-sided 95% CI | 92.87 [91.24 to NA] — One-sided 95% CI | 98.72 [98.49 to NA] — One-sided 95% CI | 95.35 [94.14 to NA] — One-sided 95% CI | 95.65 [94.74 to NA] — One-sided 95% CI

2. Secondary Outcome: Inhibition of Serum TXB2 on Days 7, 16, 17, and 19 of the In-house Treatment Period at 1, 3, 6, 12, 18, and 24 Hours (Except at 24 Hours on Day 16) Post IR ASA 81 mg Administration
Description: Inhibition of serum TXB2 at each time point were calculated using the percentage of reduction from baseline as follows: Inhibition (%) = 100 × (Baseline Value - Post-baseline Value) / Baseline Value. For primary analysis, the mean and the lower bound of the corresponding one-sided 95% CI were calculated.
Time Frame: At 1, 3, 6, 12, 18, and 24 hours on Days 7, 16, 17, and 19 (except 24 hours on Day 16)
Population: Percentages are based on the number of participants in the Evaluable Population in each treatment group.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 10 | 15
percentage
  Day 7 at 1 hour | 99.86 [99.82 to NA] — One-sided 95% CI | 99.83 [99.81 to NA] — One-sided 95% CI | 99.69 [99.63 to NA] — One-sided 95% CI | 99.67 [99.60 to NA] — One-sided 95% CI | 99.91 [99.87 to NA] — One-sided 95% CI | 99.84 [99.81 to NA] — One-sided 95% CI
  Day 7 at 3 hour | 99.84 [99.79 to NA] — One-sided 95% CI | 99.79 [99.76 to NA] — One-sided 95% CI | 99.54 [99.46 to NA] — One-sided 95% CI | 99.66 [99.58 to NA] — One-sided 95% CI | 99.86 [99.81 to NA] — One-sided 95% CI | 99.80 [99.77 to NA] — One-sided 95% CI
  Day 7 at 6 hour | 99.69 [99.58 to NA] — One-sided 95% CI | 99.67 [99.60 to NA] — One-sided 95% CI | 99.44 [99.34 to NA] — One-sided 95% CI | 99.48 [99.36 to NA] — One-sided 95% CI | 99.75 [99.63 to NA] — One-sided 95% CI | 99.70 [99.65 to NA] — One-sided 95% CI
  Day 7 at 12 hour | 99.59 [99.46 to NA] — One-sided 95% CI | 99.48 [99.42 to NA] — One-sided 95% CI | 99.12 [98.98 to NA] — One-sided 95% CI | 99.31 [99.17 to NA] — One-sided 95% CI | 99.68 [99.57 to NA] — One-sided 95% CI | 99.63 [99.56 to NA] — One-sided 95% CI
  Day 7 at 18 hour | 99.18 [99.01 to NA] — One-sided 95% CI | 99.18 [99.04 to NA] — One-sided 95% CI | 99.76 [99.71 to NA] — One-sided 95% CI | 98.86 [98.68 to NA] — One-sided 95% CI | 99.39 [99.19 to NA] — One-sided 95% CI | 99.70 [99.64 to NA] — One-sided 95% CI
  Day 7 at 24 hour | 99.01 [98.76 to NA] — One-sided 95% CI | 99.55 [99.43 to NA] — One-sided 95% CI | 97.78 [96.51 to NA] — One-sided 95% CI | 98.71 [98.46 to NA] — One-sided 95% CI | 99.23 [99.00 to NA] — One-sided 95% CI | 99.80 [99.75 to NA] — One-sided 95% CI
  Day 16 at 1 hour | 99.06 [98.79 to NA] — One-sided 95% CI | 98.38 [98.10 to NA] — One-sided 95% CI | 98.32 [98.09 to NA] — One-sided 95% CI | 99.71 [99.64 to NA] — One-sided 95% CI | 99.28 [99.08 to NA] — One-sided 95% CI | 98.81 [98.59 to NA] — One-sided 95% CI
  Day 16 at 3 hour | 98.80 [98.49 to NA] — One-sided 95% CI | 97.67 [97.41 to NA] — One-sided 95% CI | 98.02 [97.68 to NA] — One-sided 95% CI | 99.68 [99.60 to NA] — One-sided 95% CI | 99.19 [99.00 to NA] — One-sided 95% CI | 98.53 [98.23 to NA] — One-sided 95% CI
  Day 16 at 6 hour | 97.69 [97.21 to NA] — One-sided 95% CI | 96.26 [95.70 to NA] — One-sided 95% CI | 97.40 [97.03 to NA] — One-sided 95% CI | 99.55 [99.45 to NA] — One-sided 95% CI | 98.43 [98.05 to NA] — One-sided 95% CI | 97.51 [97.10 to NA] — One-sided 95% CI
  Day 16 at 12 hour | 96.59 [95.67 to NA] — One-sided 95% CI | 92.71 [91.13 to NA] — One-sided 95% CI | 96.31 [95.68 to NA] — One-sided 95% CI | 99.42 [99.29 to NA] — One-sided 95% CI | 97.84 [97.10 to NA] — One-sided 95% CI | 95.38 [94.13 to NA] — One-sided 95% CI
  Day 16 at 18 hour | 94.19 [93.04 to NA] — One-sided 95% CI | 92.23 [90.24 to NA] — One-sided 95% CI | 95.68 [94.62 to NA] — One-sided 95% CI | 99.01 [98.85 to NA] — One-sided 95% CI | 96.45 [95.43 to NA] — One-sided 95% CI | 97.73 [97.28 to NA] — One-sided 95% CI
  Day 17 at 1 hour | 95.71 [94.31 to NA] — One-sided 95% CI | 94.63 [93.66 to NA] — One-sided 95% CI | 95.56 [94.69 to NA] — One-sided 95% CI | 99.70 [99.64 to NA] — One-sided 95% CI | 97.42 [96.88 to NA] — One-sided 95% CI | 96.95 [96.30 to NA] — One-sided 95% CI
  Day 17 at 3 hour | 95.49 [94.38 to NA] — One-sided 95% CI | 92.79 [91.36 to NA] — One-sided 95% CI | 96.43 [95.89 to NA] — One-sided 95% CI | 99.68 [99.60 to NA] — One-sided 95% CI | 96.96 [96.33 to NA] — One-sided 95% CI | 95.92 [95.03 to NA] — One-sided 95% CI
  Day 17 at 6 hour | 93.55 [91.86 to NA] — One-sided 95% CI | 90.91 [89.21 to NA] — One-sided 95% CI | 95.64 [94.92 to NA] — One-sided 95% CI | 99.52 [99.41 to NA] — One-sided 95% CI | 95.31 [94.32 to NA] — One-sided 95% CI | 93.91 [92.61 to NA] — One-sided 95% CI
  Day 17 at 12 hour | 92.54 [91.08 to NA] — One-sided 95% CI | 91.15 [89.80 to NA] — One-sided 95% CI | 94.13 [93.08 to NA] — One-sided 95% CI | 99.30 [99.13 to NA] — One-sided 95% CI | 94.74 [93.62 to NA] — One-sided 95% CI | 92.60 [90.92 to NA] — One-sided 95% CI
  Day 17 at 18 hour | 89.44 [87.48 to NA] — One-sided 95% CI | 87.19 [85.43 to NA] — One-sided 95% CI | 94.23 [93.42 to NA] — One-sided 95% CI | 98.95 [98.76 to NA] — One-sided 95% CI | 93.42 [92.27 to NA] — One-sided 95% CI | 88.14 [85.42 to NA] — One-sided 95% CI
  Day 17 at 24 hour | 89.05 [86.86 to NA] — One-sided 95% CI | 83.67 [81.77 to NA] — One-sided 95% CI | 90.39 [88.57 to NA] — One-sided 95% CI | 98.70 [98.48 to NA] — One-sided 95% CI | 91.40 [89.21 to NA] — One-sided 95% CI | 84.27 [80.66 to NA] — One-sided 95% CI
  Day 19 at 1 hour | 98.35 [97.86 to NA] — One-sided 95% CI | 97.89 [97.45 to NA] — One-sided 95% CI | 98.89 [98.64 to NA] — One-sided 95% CI | 99.69 [99.62 to NA] — One-sided 95% CI | 98.16 [97.74 to NA] — One-sided 95% CI | 94.06 [92.59 to NA] — One-sided 95% CI
  Day 19 at 3 hour | 98.52 [98.02 to NA] — One-sided 95% CI | 97.90 [97.46 to NA] — One-sided 95% CI | 99.05 [98.93 to NA] — One-sided 95% CI | 99.64 [99.55 to NA] — One-sided 95% CI | 98.27 [97.92 to NA] — One-sided 95% CI | 94.44 [92.92 to NA] — One-sided 95% CI
  Day 19 at 6 hour | 98.26 [97.78 to NA] — One-sided 95% CI | 97.43 [96.73 to NA] — One-sided 95% CI | 98.98 [98.81 to NA] — One-sided 95% CI | 99.50 [99.39 to NA] — One-sided 95% CI | 97.84 [97.34 to NA] — One-sided 95% CI | 93.25 [91.11 to NA] — One-sided 95% CI
  Day 19 at 12 hour | 97.67 [96.95 to NA] — One-sided 95% CI | 96.90 [96.06 to NA] — One-sided 95% CI | 98.77 [98.57 to NA] — One-sided 95% CI | 99.26 [99.09 to NA] — One-sided 95% CI | 97.33 [96.70 to NA] — One-sided 95% CI | 92.00 [89.44 to NA] — One-sided 95% CI
  Day 19 at 18 hour | 97.21 [96.40 to NA] — One-sided 95% CI | 96.29 [95.40 to NA] — One-sided 95% CI | 98.52 [98.27 to NA] — One-sided 95% CI | 98.88 [98.67 to NA] — One-sided 95% CI | 96.62 [95.86 to NA] — One-sided 95% CI | 90.94 [88.41 to NA] — One-sided 95% CI
  Day 19 at 24 hour | 97.04 [96.13 to NA] — One-sided 95% CI | 96.16 [95.25 to NA] — One-sided 95% CI | 97.98 [97.72 to NA] — One-sided 95% CI | 98.49 [98.19 to NA] — One-sided 95% CI | 96.01 [94.86 to NA] — One-sided 95% CI | 90.67 [88.25 to NA] — One-sided 95% CI

3. Secondary Outcome: Inhibition of Arachidonic Acid (AA)-Induced Platelet Aggregation on Days 7, 16, 17, and 19 at 1, 3, 6, 12, 18, and 24 Hours Post IR ASA 81 mg Administration
Description: Inhibition of AA-induced platelet aggregation at each time point were calculated using the percentage of reduction from baseline as follows: Inhibition (%) = 100 × (Baseline Value - Post-baseline Value) / Baseline Value. For primary analysis, the mean and the lower bound of the corresponding one-sided 95% CI were calculated. The platelet aggregation change-from-baseline scores range broadly in large part due to inclusion of participants with low baseline platelet aggregation scores.
Time Frame: At 1, 3, 6, 12, 18, and 24 hours on Days 7, 16, 17, and 19
Population: Percentages are based on the number of participants in the Evaluable Population in each treatment group. Evaluable participants number in Group 4 at time point Day 7/1 Hour was 12; 11 in group 6, 7 in Group 5, 12 in Group 6 at Day 16/1 Hour.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 10 | 14
percentage
  Day 7 at 1 hour | 58.60 (58.893) [29.49 to NA] — One-sided 95% CI | 12.78 (139.818) [-53.40 to NA] — One-sided 95% CI | 5.55 (306.389) [-133.79 to NA] — One-sided 95% CI | 87.73 (8.777) [83.18 to NA] — One-sided 95% CI | 64.14 (40.389) [40.73 to NA] — One-sided 95% CI | 30.45 (182.916) [-56.12 to NA] — One-sided 95% CI
  Day 7 at 3 hour | -121.76 (630.765) [-433.56 to NA] — One-sided 95% CI | 12.86 (144.823) [-55.68 to NA] — One-sided 95% CI | 10.80 (280.405) [-116.72 to NA] — One-sided 95% CI | 79.16 (29.318) [64.67 to NA] — One-sided 95% CI | 75.89 (24.067) [61.94 to NA] — One-sided 95% CI | 18.99 (222.208) [-86.18 to NA] — One-sided 95% CI
  Day 7 at 6 hour | 61.74 (63.400) [30.40 to NA] — One-sided 95% CI | 1.70 (168.415) [-78.01 to NA] — One-sided 95% CI | -3.29 (331.881) [-154.22 to NA] — One-sided 95% CI | 78.20 (33.051) [61.86 to NA] — One-sided 95% CI | 73.69 (31.859) [55.22 to NA] — One-sided 95% CI | 26.91 (183.636) [-60.00 to NA] — One-sided 95% CI
  Day 7 at 12 hour | 36.41 (162.350) [-43.85 to NA] — One-sided 95% CI | 28.54 (113.063) [-24.98 to NA] — One-sided 95% CI | -17.95 (275.811) [-143.38 to NA] — One-sided 95% CI | 80.81 (33.244) [64.37 to NA] — One-sided 95% CI | 76.02 (26.733) [60.52 to NA] — One-sided 95% CI | 17.11 (249.918) [-101.18 to NA] — One-sided 95% CI
  Day 7 at 18 hour | 62.36 (68.382) [28.56 to NA] — One-sided 95% CI | 25.27 (119.755) [-31.41 to NA] — One-sided 95% CI | 11.96 (280.718) [-115.70 to NA] — One-sided 95% CI | 78.50 (37.671) [59.88 to NA] — One-sided 95% CI | 38.58 (138.715) [-41.83 to NA] — One-sided 95% CI | -151.06 (863.434) [-559.72 to NA] — One-sided 95% CI
  Day 7 at 24 hour | 80.60 (26.517) [67.50 to NA] — One-sided 95% CI | 46.31 (91.924) [2.80 to NA] — One-sided 95% CI | 41.29 (178.089) [-39.70 to NA] — One-sided 95% CI | 89.12 (18.535) [79.96 to NA] — One-sided 95% CI | 77.61 (29.401) [60.57 to NA] — One-sided 95% CI | 44.02 (157.466) [-30.51 to NA] — One-sided 95% CI
  Day 16 at 1 hour | 68.96 (39.662) [49.36 to NA] — One-sided 95% CI | 24.15 (114.782) [-38.58 to NA] — One-sided 95% CI | 29.25 (229.744) [-75.23 to NA] — One-sided 95% CI | 86.12 (21.728) [75.38 to NA] — One-sided 95% CI | 62.67 (45.474) [29.27 to NA] — One-sided 95% CI | 45.12 (141.196) [-28.08 to NA] — One-sided 95% CI
  Day 16 at 3 hour | 75.25 (42.568) [54.21 to NA] — One-sided 95% CI | 51.22 (74.825) [15.81 to NA] — One-sided 95% CI | 33.12 (203.704) [-59.52 to NA] — One-sided 95% CI | 85.92 (21.762) [75.16 to NA] — One-sided 95% CI | 83.51 (21.986) [70.77 to NA] — One-sided 95% CI | 37.09 (170.694) [-43.70 to NA] — One-sided 95% CI
  Day 16 at 6 hour | 74.45 (42.678) [53.35 to NA] — One-sided 95% CI | 61.20 (63.333) [31.22 to NA] — One-sided 95% CI | 62.32 (100.840) [16.46 to NA] — One-sided 95% CI | 81.36 (37.422) [62.86 to NA] — One-sided 95% CI | 82.55 (17.893) [72.18 to NA] — One-sided 95% CI | 81.07 (26.570) [68.49 to NA] — One-sided 95% CI
  Day 16 at 12 hour | 79.88 (26.425) [66.81 to NA] — One-sided 95% CI | 70.98 (51.499) [46.61 to NA] — One-sided 95% CI | 11.16 (254.042) [-104.37 to NA] — One-sided 95% CI | 81.38 (31.472) [65.82 to NA] — One-sided 95% CI | 79.51 (21.218) [67.21 to NA] — One-sided 95% CI | 53.04 (118.315) [-2.96 to NA] — One-sided 95% CI
  Day 16 at 18 hour | 73.86 (36.769) [55.68 to NA] — One-sided 95% CI | 74.07 (40.473) [54.92 to NA] — One-sided 95% CI | 35.43 (204.054) [-57.37 to NA] — One-sided 95% CI | 85.19 (25.762) [72.45 to NA] — One-sided 95% CI | 71.93 (52.602) [41.44 to NA] — One-sided 95% CI | 71.64 (52.123) [46.97 to NA] — One-sided 95% CI
  Day 16 at 24 hour | 67.47 (37.467) [48.95 to NA] — One-sided 95% CI | 64.26 (51.050) [40.10 to NA] — One-sided 95% CI | 15.96 (281.846) [-112.22 to NA] — One-sided 95% CI | 85.25 (18.848) [75.93 to NA] — One-sided 95% CI | 73.73 (32.648) [54.81 to NA] — One-sided 95% CI | 51.40 (116.489) [-3.73 to NA] — One-sided 95% CI
  Day 17 at 1 hour | 76.23 (30.966) [60.92 to NA] — One-sided 95% CI | 56.77 (63.792) [26.57 to NA] — One-sided 95% CI | -452.48 (2088.027) [-1402.05 to NA] — One-sided 95% CI | 83.53 (25.476) [70.94 to NA] — One-sided 95% CI | 82.13 (19.364) [70.90 to NA] — One-sided 95% CI | 33.64 (197.114) [-59.65 to NA] — One-sided 95% CI
  Day 17 at 3 hour | 78.48 (27.969) [64.66 to NA] — One-sided 95% CI | 46.16 (79.122) [8.71 to NA] — One-sided 95% CI | 21.74 (255.742) [-94.56 to NA] — One-sided 95% CI | 83.48 (25.466) [70.89 to NA] — One-sided 95% CI | 75.15 (30.948) [57.21 to NA] — One-sided 95% CI | 48.27 (117.511) [-7.35 to NA] — One-sided 95% CI
  Day 17 at 6 hour | 76.46 (36.017) [58.65 to NA] — One-sided 95% CI | 69.16 (43.503) [48.57 to NA] — One-sided 95% CI | 37.52 (204.341) [-55.41 to NA] — One-sided 95% CI | 83.48 (25.514) [70.87 to NA] — One-sided 95% CI | 74.61 (38.546) [52.27 to NA] — One-sided 95% CI | 52.03 (131.415) [-10.17 to NA] — One-sided 95% CI
  Day 17 at 12 hour | 83.17 (20.398) [73.08 to NA] — One-sided 95% CI | 86.40 (17.991) [77.88 to NA] — One-sided 95% CI | -24.72 (408.994) [-210.72 to NA] — One-sided 95% CI | 86.00 (17.935) [77.13 to NA] — One-sided 95% CI | 82.37 (27.172) [66.62 to NA] — One-sided 95% CI | 67.55 (79.461) [29.95 to NA] — One-sided 95% CI
  Day 17 at 18 hour | 82.30 (22.570) [71.15 to NA] — One-sided 95% CI | 68.65 (45.824) [46.96 to NA] — One-sided 95% CI | 31.96 (178.297) [-49.12 to NA] — One-sided 95% CI | 83.71 (25.383) [71.17 to NA] — One-sided 95% CI | 71.35 (31.709) [52.97 to NA] — One-sided 95% CI | 41.51 (144.334) [-26.81 to NA] — One-sided 95% CI
  Day 17 at 24 hour | 78.66 (36.988) [60.37 to NA] — One-sided 95% CI | 70.84 (46.622) [48.77 to NA] — One-sided 95% CI | 53.24 (103.247) [6.29 to NA] — One-sided 95% CI | 85.43 (25.873) [72.64 to NA] — One-sided 95% CI | 82.13 (29.286) [65.15 to NA] — One-sided 95% CI | 87.02 (23.703) [75.80 to NA] — One-sided 95% CI
  Day 19 at 1 hour | 64.06 (64.304) [32.28 to NA] — One-sided 95% CI | 41.10 (103.816) [-8.04 to NA] — One-sided 95% CI | 21.46 (255.470) [-94.72 to NA] — One-sided 95% CI | 83.97 (25.386) [71.42 to NA] — One-sided 95% CI | 81.05 (19.743) [69.60 to NA] — One-sided 95% CI | 43.92 (157.676) [-30.71 to NA] — One-sided 95% CI
  Day 19 at 3 hour | 69.18 (58.761) [40.13 to NA] — One-sided 95% CI | 48.51 (73.341) [13.80 to NA] — One-sided 95% CI | 23.64 (228.479) [-80.27 to NA] — One-sided 95% CI | 81.62 (33.415) [65.10 to NA] — One-sided 95% CI | 78.01 (26.265) [62.78 to NA] — One-sided 95% CI | 14.85 (263.930) [-110.07 to NA] — One-sided 95% CI
  Day 19 at 6 hour | 60.96 (72.629) [25.06 to NA] — One-sided 95% CI | 50.21 (77.242) [13.65 to NA] — One-sided 95% CI | 51.59 (126.753) [-6.05 to NA] — One-sided 95% CI | 82.98 (29.512) [68.39 to NA] — One-sided 95% CI | 70.87 (35.515) [50.28 to NA] — One-sided 95% CI | 58.64 (105.239) [8.83 to NA] — One-sided 95% CI
  Day 19 at 12 hour | 1.08 (313.927) [-154.10 to NA] — One-sided 95% CI | 33.43 (110.105) [-18.68 to NA] — One-sided 95% CI | 36.92 (204.360) [-56.02 to NA] — One-sided 95% CI | 84.45 (25.743) [71.72 to NA] — One-sided 95% CI | 44.97 (112.099) [-20.01 to NA] — One-sided 95% CI | 13.17 (215.066) [-88.62 to NA] — One-sided 95% CI
  Day 19 at 18 hour | 69.69 (57.918) [41.06 to NA] — One-sided 95% CI | 74.55 (46.130) [52.71 to NA] — One-sided 95% CI | 15.41 (281.253) [-112.49 to NA] — One-sided 95% CI | 91.12 (4.541) [88.88 to NA] — One-sided 95% CI | 88.43 (10.953) [82.08 to NA] — One-sided 95% CI | 84.46 (28.685) [70.88 to NA] — One-sided 95% CI
  Day 19 at 24 hour | 89.86 (13.568) [83.15 to NA] — One-sided 95% CI | 80.90 (28.329) [67.49 to NA] — One-sided 95% CI | 29.02 (230.055) [-75.60 to NA] — One-sided 95% CI | 83.67 (34.194) [66.77 to NA] — One-sided 95% CI | 82.63 (20.393) [70.80 to NA] — One-sided 95% CI | 71.27 (57.042) [44.27 to NA] — One-sided 95% CI

4. Secondary Outcome: Inhibition of TXB2 Using Platelet-rich Plasma (PRP) on Days 7, 16, 17, and 19 of the In-house Treatment Period at 1, 3, 6, 12, 18, and 24 Hours Post IR ASA 81 mg Administration
Description: Inhibition of plasma TXB2 at each time point were calculated using the percentage of reduction from baseline as follows: Inhibition (%) = 100 × (Baseline Value - Post-baseline Value) / Baseline Value. For primary analysis, the mean and the lower bound of the corresponding one-sided 95% CI were calculated.
Time Frame: At 1, 3, 6, 12, 18, and 24 hours on Days 7, 16, 17, and 19
Population: Percentages are based on the number of participants in the Evaluable Population in each treatment group. Evaluable participants number in Group 1 at time point Day 7/1 Hour, Day 7/3 Hour, Day 7/6 Hour, Day 7/12 Hour was 12.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 10 | 15
percentage
  Day 7 at 1 hour | 98.84 [98.35 to NA] — One-sided 95% CI | 98.82 [98.33 to NA] — One-sided 95% CI | 97.59 [96.62 to NA] — One-sided 95% CI | 98.34 [97.61 to NA] — One-sided 95% CI | 99.40 [99.17 to NA] — One-sided 95% CI | 98.67 [98.14 to NA] — One-sided 95% CI
  Day 7 at 3 hour | 97.82 [97.00 to NA] — One-sided 95% CI | 98.25 [97.48 to NA] — One-sided 95% CI | 97.72 [97.03 to NA] — One-sided 95% CI | 97.61 [96.55 to NA] — One-sided 95% CI | 98.95 [98.49 to NA] — One-sided 95% CI | 97.68 [96.44 to NA] — One-sided 95% CI
  Day 7 at 6 hour | 97.95 [96.59 to NA] — One-sided 95% CI | 98.57 [97.83 to NA] — One-sided 95% CI | 98.37 [97.63 to NA] — One-sided 95% CI | 97.29 [96.46 to NA] — One-sided 95% CI | 99.06 [98.42 to NA] — One-sided 95% CI | 97.93 [97.29 to NA] — One-sided 95% CI
  Day 7 at 12 hour | 97.75 [96.69 to NA] — One-sided 95% CI | 97.92 [96.72 to NA] — One-sided 95% CI | 96.66 [95.59 to NA] — One-sided 95% CI | 97.49 [96.71 to NA] — One-sided 95% CI | 98.54 [97.70 to NA] — One-sided 95% CI | 98.36 [97.52 to NA] — One-sided 95% CI
  Day 7 at 18 hour | 97.85 [96.65 to NA] — One-sided 95% CI | 96.09 [94.63 to NA] — One-sided 95% CI | 98.79 [98.32 to NA] — One-sided 95% CI | 96.29 [94.83 to NA] — One-sided 95% CI | 97.97 [96.94 to NA] — One-sided 95% CI | 97.87 [96.98 to NA] — One-sided 95% CI
  Day 7 at 24 hour | 96.62 [95.38 to NA] — One-sided 95% CI | 98.26 [97.59 to NA] — One-sided 95% CI | 98.89 [98.42 to NA] — One-sided 95% CI | 95.04 [93.35 to NA] — One-sided 95% CI | 98.13 [97.54 to NA] — One-sided 95% CI | 98.44 [97.81 to NA] — One-sided 95% CI
  Day 16 at 1 hour | 98.06 [97.15 to NA] — One-sided 95% CI | 95.49 [93.79 to NA] — One-sided 95% CI | 89.55 [87.09 to NA] — One-sided 95% CI | 98.99 [98.59 to NA] — One-sided 95% CI | 96.73 [95.54 to NA] — One-sided 95% CI | 94.95 [92.99 to NA] — One-sided 95% CI
  Day 16 at 3 hour | 93.03 [90.35 to NA] — One-sided 95% CI | 89.25 [85.98 to NA] — One-sided 95% CI | 92.62 [90.24 to NA] — One-sided 95% CI | 97.37 [96.45 to NA] — One-sided 95% CI | 96.17 [95.16 to NA] — One-sided 95% CI | 90.62 [87.59 to NA] — One-sided 95% CI
  Day 16 at 6 hour | 93.55 [89.83 to NA] — One-sided 95% CI | 88.62 [83.96 to NA] — One-sided 95% CI | 90.40 [88.30 to NA] — One-sided 95% CI | 98.50 [97.89 to NA] — One-sided 95% CI | 95.56 [93.74 to NA] — One-sided 95% CI | 91.27 [87.89 to NA] — One-sided 95% CI
  Day 16 at 12 hour | 89.55 [86.80 to NA] — One-sided 95% CI | 85.63 [80.50 to NA] — One-sided 95% CI | 88.76 [85.89 to NA] — One-sided 95% CI | 97.42 [96.77 to NA] — One-sided 95% CI | 92.30 [90.55 to NA] — One-sided 95% CI | 89.45 [84.52 to NA] — One-sided 95% CI
  Day 16 at 18 hour | 86.61 [82.69 to NA] — One-sided 95% CI | 84.41 [80.03 to NA] — One-sided 95% CI | 82.14 [75.75 to NA] — One-sided 95% CI | 95.69 [94.57 to NA] — One-sided 95% CI | 93.28 [91.00 to NA] — One-sided 95% CI | 91.03 [87.81 to NA] — One-sided 95% CI
  Day 16 at 24 hour | 86.42 [80.81 to NA] — One-sided 95% CI | 72.66 [65.53 to NA] — One-sided 95% CI | 77.71 [72.15 to NA] — One-sided 95% CI | 95.78 [94.35 to NA] — One-sided 95% CI | 88.49 [84.08 to NA] — One-sided 95% CI | 86.87 [81.86 to NA] — One-sided 95% CI
  Day 17 at 1 hour | 86.19 [80.48 to NA] — One-sided 95% CI | 79.99 [74.59 to NA] — One-sided 95% CI | 86.14 [83.15 to NA] — One-sided 95% CI | 98.72 [98.30 to NA] — One-sided 95% CI | 93.75 [91.26 to NA] — One-sided 95% CI | 90.00 [84.47 to NA] — One-sided 95% CI
  Day 17 at 3 hour | 85.45 [79.85 to NA] — One-sided 95% CI | 90.16 [87.39 to NA] — One-sided 95% CI | 92.60 [90.38 to NA] — One-sided 95% CI | 98.01 [97.13 to NA] — One-sided 95% CI | 88.52 [84.47 to NA] — One-sided 95% CI | 83.94 [78.25 to NA] — One-sided 95% CI
  Day 17 at 6 hour | 82.90 [75.87 to NA] — One-sided 95% CI | 84.77 [80.99 to NA] — One-sided 95% CI | 83.08 [77.53 to NA] — One-sided 95% CI | 97.34 [96.57 to NA] — One-sided 95% CI | 92.39 [89.45 to NA] — One-sided 95% CI | 85.82 [79.55 to NA] — One-sided 95% CI
  Day 17 at 12 hour | 83.49 [76.38 to NA] — One-sided 95% CI | 81.22 [75.88 to NA] — One-sided 95% CI | 86.50 [82.09 to NA] — One-sided 95% CI | 97.46 [96.40 to NA] — One-sided 95% CI | 92.42 [88.90 to NA] — One-sided 95% CI | 82.13 [76.07 to NA] — One-sided 95% CI
  Day 17 at 18 hour | 85.77 [81.67 to NA] — One-sided 95% CI | 78.34 [72.79 to NA] — One-sided 95% CI | 86.53 [82.83 to NA] — One-sided 95% CI | 95.47 [93.79 to NA] — One-sided 95% CI | 85.70 [82.50 to NA] — One-sided 95% CI | 70.90 [62.89 to NA] — One-sided 95% CI
  Day 17 at 24 hour | 79.55 [72.74 to NA] — One-sided 95% CI | 79.06 [72.89 to NA] — One-sided 95% CI | 75.67 [70.44 to NA] — One-sided 95% CI | 97.23 [96.19 to NA] — One-sided 95% CI | 92.07 [89.87 to NA] — One-sided 95% CI | 81.34 [76.55 to NA] — One-sided 95% CI
  Day 19 at 1 hour | 92.68 [89.50 to NA] — One-sided 95% CI | 89.65 [86.17 to NA] — One-sided 95% CI | 95.32 [93.74 to NA] — One-sided 95% CI | 98.05 [97.37 to NA] — One-sided 95% CI | 94.39 [91.69 to NA] — One-sided 95% CI | 79.36 [73.75 to NA] — One-sided 95% CI
  Day 19 at 3 hour | 91.03 [88.18 to NA] — One-sided 95% CI | 92.04 [90.13 to NA] — One-sided 95% CI | 93.68 [91.71 to NA] — One-sided 95% CI | 97.82 [97.16 to NA] — One-sided 95% CI | 94.53 [91.78 to NA] — One-sided 95% CI | 79.82 [74.39 to NA] — One-sided 95% CI
  Day 19 at 6 hour | 90.57 [87.64 to NA] — One-sided 95% CI | 91.49 [88.95 to NA] — One-sided 95% CI | 92.35 [90.34 to NA] — One-sided 95% CI | 98.24 [97.66 to NA] — One-sided 95% CI | 93.72 [90.55 to NA] — One-sided 95% CI | 81.14 [77.02 to NA] — One-sided 95% CI
  Day 19 at 12 hour | 91.59 [88.31 to NA] — One-sided 95% CI | 89.25 [86.51 to NA] — One-sided 95% CI | 95.18 [93.46 to NA] — One-sided 95% CI | 96.91 [95.87 to NA] — One-sided 95% CI | 92.84 [90.52 to NA] — One-sided 95% CI | 80.66 [75.32 to NA] — One-sided 95% CI
  Day 19 at 18 hour | 91.20 [87.58 to NA] — One-sided 95% CI | 93.50 [91.00 to NA] — One-sided 95% CI | 94.85 [92.96 to NA] — One-sided 95% CI | 96.24 [95.27 to NA] — One-sided 95% CI | 92.74 [89.92 to NA] — One-sided 95% CI | 85.67 [81.17 to NA] — One-sided 95% CI
  Day 19 at 24 hour | 93.76 [91.18 to NA] — One-sided 95% CI | 90.93 [87.80 to NA] — One-sided 95% CI | 93.66 [91.58 to NA] — One-sided 95% CI | 96.63 [95.39 to NA] — One-sided 95% CI | 96.14 [93.74 to NA] — One-sided 95% CI | 81.67 [74.94 to NA] — One-sided 95% CI

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected after first dose of investigational product on Day 1 until completion of all study procedures throughout the study.
Description: Tables represent all adverse events in the Safety Population (all randomized participants who took at least 1 dose of investigational product) during the aspirin mono-therapy run-in phase, the treatment phase and the aspirin mono-therapy run-out phase.
Groups:
- Group 0-IR ASA 81 mg qd in Run-in Period: Participants, subsequently randomized to treatment period, were administered the first dose of immediate release acetylsalicylic acid (IR ASA, Aspirin, BAYE4465) 81 mg once daily at the clinical study site and instructed to take the remaining 5 doses in a fasted state with a full glass of water once daily in the morning in an outpatient setting.
Arm/Group | Group 0-IR ASA 81 mg qd in Run-in Period | Group 1-IR ASA Co-administered With Naproxen Sodium | Group 2-IR ASA 30 Min After Naproxen Sodium | Group 3-IR ASA 8 Hours After Naproxen Sodium | Group 4-IR ASA Only | Group 5-IR ASA 30 Min Before Naproxen Sodium | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/102 | 4/17 | 1/17 | 4/17 | 3/17 | 2/17 | 4/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 0-IR ASA 81 mg qd in Run-in Period (N=102) | Group 1-IR ASA Co-administered With Naproxen Sodium (N=17) | Group 2-IR ASA 30 Min After Naproxen Sodium (N=17) | Group 3-IR ASA 8 Hours After Naproxen Sodium (N=17) | Group 4-IR ASA Only (N=17) | Group 5-IR ASA 30 Min Before Naproxen Sodium (N=17) | Group 6-IR ASA 30 Min After First Dose of Naproxen Sodium Bid (N=17)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coagulation time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other